CLINICAL TRIAL: NCT03286192
Title: Compassion Cultivation Training for Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Debbie Anglade, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20170290
Record Dates: First submitted 2017-09-05; First posted 2017-09-18 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Feasibility

STUDY DESIGN:
Intervention Model Description: Single group feasibility study of a psychosocial intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Intervention (Experimental): All participants in this arm receive compassion cultivation training
  Interventions: Behavioral: compassion cultivation training

INTERVENTIONS:
Behavioral: compassion cultivation training — Eight 2-hour group sessions that provide a structured and systematic way of cultivating daily-life skills needed to strengthen qualities of compassion, empathy, and kindness for oneself and others.

SUMMARY:
The purpose of this study is to evaluate the feasibility of implementing a Compassion Cultivation Training (CCT) program for oncology nurses at Sylvester Comprehensive Cancer Center. The goal of CCT is to provide a structured and systematic way of cultivating daily-life skills needed to strengthen qualities of compassion, empathy, and kindness for oneself and others. CCT typically includes (i) eight weekly 2-hour classes and (ii) daily practice. The in-class activities include pedagogical instruction and active group discussion, guided meditation, interactive practical exercises, and sharing of inspiring readings/stories to prime feelings of open-heartedness or connection to others.

DETAILED DESCRIPTION:
The Compassion Cultivation Training (CCT) protocol is a secular course that was developed by the Center for Compassion & Altruism Research and Education (CCARE) at Stanford University, School of Medicine (Jinpa, 2013). The course was developed by Thupten Jinpa, PhD, in collaboration with contemplative scholars, psychologists, and scientist at Stanford. The goal of CCT is to provide a structured and systematic way of cultivating daily-life skills needed to strengthen qualities of compassion, empathy, and kindness for oneself and others. CCT typically includes (i) eight weekly 2-hour classes and (ii) daily practice. The in-class activities include pedagogical instruction and active group discussion, guided meditation, interactive practical exercises, and sharing of inspiring readings/stories to prime feelings of open-heartedness or connection to others. The daily practice includes both formal and informal practices. Participants are provided with formal guided meditations that are 15 to 30 minutes long in the form of MP3 or cds. Participants may receive practices and instructions via email with a link to the location of the MP3. They will be provided with practice logs to report their amount of practice as well as some basic observations to the research team. In the present study, we will follow the official CCT manual. The training is composed of 8 sessions, which can be delivered in 7-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older
2. Be willing and able to give informed consent
3. Be a Registered Nurse (RN)
4. Currently works at Sylvester Comprehensive Cancer Center
5. Currently works at least 20 hours/week
6. Be able to speak and read English

Exclusion Criteria:

1. Any participants who are deemed to present an acute safety risk to self or others.
2. Any infants, children, or teenagers under 18 years of age.
3. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Number of individuals who do not drop out of the study prior to completing the post-intervention assessment | 24 weeks after first session
  Number of individuals who do not drop out of the study prior to completing the post-intervention assessment

SECONDARY OUTCOMES:
Perceived Stress Scale | baseline and 7-10 weeks
  self-report instrument that measures perceptions of stress
Maslach Burnout Inventory | baseline and 7-10 weeks
  self-report instrument that measures emotional exhaustion, depersonalization, and acheivement
Philadelphia Mindfulness Scale | baseline and 7-10 weeks
  self-report instrument that measures present moment awareness and acceptance
Distress Tolerance Scale | baseline and 7-10 weeks
  self-report instrument that measures feelings of distress
SF-36 | baseline and 7-10 weeks
  self-report measure of health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Anglade, PhD, Principal Investigator — University of Miami
Locations (1):
- Sylvester Comprehensive Cancer Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03286192/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03286192/Prot_SAP_002.pdf